CLINICAL TRIAL: NCT04335461
Title: Postoperative Pain Control in Extracapsular Hip Fracture Patients: Fascia Iliaca Compartment Block Versus Fracture Block
Brief Title: Postop Pain Control in Hip Fracture Surgery: Fascia Iliaca Compartment Block Versus Fracture Block
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn. Study expired in IRB system and no patients enrolled as per institutional CTMS and IRB systems. Primary and Study Completion Dates reflect date IRB approval expired.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-10737
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hip Fractures; Analgesia; Opioid Use; Pain, Postoperative
MeSH Terms: conditions — Hip Fractures; Agnosia; Pain, Postoperative | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will occur at time of enrollment using unmarked envelopes. After consent, patients will be assigned a study ID that will be transcribed on the opaque envelope. The envelope will be unsealed in the operating room at time of surgery to determine the planned intervention, and it's contents will not be made available to the study personnel gathering postoperative pain data. The envelopes and randomization assignments will be kept in a locked, secured location. The only study personnel who will be unblinded are the operating surgeon and residents and physican assistants assisting in the operating room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo group, with no regional nerve blockade administered.
  Interventions: Procedure: Cephalomedullary nailing of extracapsular hip fracture; Device: cephalomedullary nail
- Fracture block (Experimental): Patients will have an intrafragmentary fracture block using fluoroscopy guidance after surgical fixation with 30cc 0.25% marcaine
  Interventions: Procedure: Cephalomedullary nailing of extracapsular hip fracture; Device: cephalomedullary nail; Drug: Regional Anesthetics
- Fascia iliaca block (Experimental): Fascia iliaca compartment blockade administered after surgical fixation using the loss of resistance technique with 30cc 0.25% marcaine
  Interventions: Procedure: Cephalomedullary nailing of extracapsular hip fracture; Device: cephalomedullary nail; Drug: Regional Anesthetics

INTERVENTIONS:
Procedure: Cephalomedullary nailing of extracapsular hip fracture — All patients will undergo cephalomedullary nailing of their extracapsular hip fractures. Both short and long nails will be used based on fracture morphology.
Device: cephalomedullary nail — Implants to be used will be variable, but include Stryker Gamma, Synthes Trochanteric Fixation Nail, Smith and Nephew Intertan.
Drug: Regional Anesthetics — Marcaine 0.25% will be administered for the two experimental arms, as described in above protocol.
  Other Names: Local anesthetics
  Arms: Fascia iliaca block; Fracture block

SUMMARY:
The investigators propose to investigate the effect of intraoperative FICB and intrafragmentary fracture blockade on postoperative pain and opiate consumption using a randomized controlled trial study design. There will be three treatment groups: (1) fascia iliaca compartment blockade administered after surgical fixation using the loss of resistance technique with 30cc 0.25% marcaine (2) intrafragmentary fracture block using fluoroscopy guidance after surgical fixation with 30cc 0.25% marcaine and (3) placebo group, with no intervention.

DETAILED DESCRIPTION:
The incidence of fragility hip fractures in elderly patients is increasing steadily in the United States and worldwide, and the mortality, morbidity and economic impact of this injury is staggering. The injury itself can result in severe pain, both preoperatively and throughout the perioperative course. These patients are also at increased risk for delirium. They are by definition elderly, and often have multiple comorbidities in addition to underlying cognitive dysfunction. Current studies estimate that the incidence of delirium after a hip fracture approaches 30%, and there is a well-established though not completely understood interaction between opioid use in elderly patients and delirium. Pain and delirium are not only poor outcomes in themselves, but they can also interfere with the rehabilitation necessary for a successful outcome after hip fracture surgery. For this reason, the topic of multimodal pain management in hip fracture patients has gained considerable traction.

One popular "opioid-sparing" strategy in these patients is regional pain blockades, administered by an anesthesia block team or by emergency room physicians. Due to the neuroanatomy of the hip region, which has sensory innervations from the sciatic, femoral, and obturator nerve, with lesser contributions from the nerve to quadratus femoris and superior gluteal nerve, effective regional blockade of the hip joint with existing methods can be a challenge. One commonly employed and researched block is the fascia iliaca compartment block (FICB), a regional block administered under ultrasound guidance or anatomical landmarks that targets the femoral nerve, the lateral femoral cutaneous nerve, and to a lesser extent, the obturator nerve. Various studies of FICB and the closely related femoral nerve block have demonstrated benefits in pain control, ease of positioning, and reduction in opiate use, and systematic reviews have concluded that the fascia iliaca compartment block is a useful and safe method to enhance preoperative pain control in hip fracture patients. However, prior research has focused on the preoperative period, with blocks placed by an anesthesia team or emergency room physicians shortly after presentation and diagnosis of a hip fracture. Additionally, no distinction is made between intracapsular or extracapsular hip fractures, except in scattered post-hoc analyses. Our project aims to investigate the efficacy of a FICB administered intraoperatively by the operating surgeon on extracapsular hip fracture patients. In addition, the investigators propose investigating intrafragmentary blockade at the fracture site itself. Fracture hematoma blocks are used extensively in orthopedics, and have demonstrated pain control equivalent to conscious sedation for the manipulation of ankle and distal radius fractures.

Study Design

The investigators propose to investigate the effect of intraoperative FICB and intrafragmentary fracture blockade on postoperative pain and opiate consumption using a randomized controlled trial study design. There will be three treatment groups: (1) fascia iliaca compartment blockade administered after surgical fixation using the loss of resistance technique with 30cc 0.25% marcaine (2) intrafragmentary fracture block using fluoroscopy guidance after surgical fixation with 30cc 0.25% marcaine and (3) placebo group, with no intervention

Randomization will occur at time of enrollment using unmarked envelopes. After consent, patients will be assigned a study ID that will be transcribed on the opaque envelope. The envelope will be unsealed in the operating room at time of surgery to determine the planned intervention, and it's contents will not be made available to the study personnel gathering postoperative pain data. The envelopes and randomization assignments will be kept in a locked, secured location. The only study personnel who will be unblinded are the operating surgeon and residents and physican assistants assisting in the operating room. Study personnel who participate in the case will not collect postoperative pain data.

The investigators will monitor various safety outcomes, including perioperative cardiac or respiratory events, mortality, and escalation of care (i.e. SICU transfer). Each adverse event will be analyzed by the senior operating surgeons to determine if the study intervention could have had a role in the event.

Our outcome measurements are pain visual analogue scores and narcotic use postoperatively. Calculations of narcotic use will be standardized to IV morphine equivalents. The associated primary and secondary hypotheses are as follows:

* Primary: There is a statistically significant difference in pain visual analogue scale (VAS) between extracapsular hip fracture patients treated intraoperatively with fascia iliaca block, fracture block, or conventional analgesia in the first 24 hours postoperatively.
* Secondary: There is a statistically significant difference in opioid consumption (measured in IV morphine equivalents / time) between extracapsular hip fracture patients treated intraoperatively with fascia iliaca block, fracture block, or conventional analgesia in the first 24 hours postoperatively.

Study Population

Our study population will be focused on elderly patients with low energy extracapsular (intertrochonteric, subtrochanteric) hip fractures. Inclusion criteria will include age 60 years or older, low energy mechanism (i.e. mechanical or syncopal fall from ground level), and extracapsular location as defined on AP and lateral radiographs of the hip. Exclusion criteria includes polytrauma patients with multiple injuries, high energy mechanisms (i.e. pedestrian struck, motor vehicle collision, fall from height), inability for the patient to consent for themselves, pathologic fracture types (secondary to tumor or atypical fractures due to bisphosphonate use), and intolerance or allergies to opioids or local anethestics.

Sample size projections target a sample of 105 patients, 35 in each group. This is based on calculation of 80% power to detect a 10mm difference in the VAS score using means and standard deviations from previous publications with measurements of pain scores in hip fracture patients. Since the duration of followup is limited to the immediate postoperative period, the investigators do not anticipate a significant drop out or loss-to-follow up rate.

Recruitment

Recruitment will occur in the emergency department by study personnel. After diagnosis of an extracapsular hip fracture is made, the exclusion and inclusion criteria will be reviewed, and eligible patients will be approached for voluntary participation in the research study.

Informed Consent

Study personnel will obtain consent in the emergency room or shortly after admission to the floor. Please find attached the planned consent form.

Risks

The proposed intervention, marcaine for regional blockade, has been studied extensively, and has been demonstrated to be safe. The risk of intravascular introduction of lidocaine is possible, but exceedingly rare. Per standarad procedure, the investigators will plan to aspirate the syringe before injection to confirm extravascular targeting. Another known risk of regional blockade is muscle weakness in the immediate postoperative period due to blockade of motor nerves. If not appropriately managed, this could create a risk of falling. Patients are routinely assessed by physical therapy for strength and muscle control before attempting ambulation postoperatively, and this will continue to be the practice. Furthermore, postoperative hip fracture patients, if they do ambulate post operative day 0, are closely assisted by physical therapists, reducing the risk of fall.

Data Analysis

Differences between study groups in regards to their baseline characteristics and outcomes will be assessed using two-sided Fisher's exact tests, chi-square tests for categorical variables, and independent samples student T-tests for continuous variables. The investigators will plan to undertake a multivariable analyses as well.

Data Quality and Management

The investigators plan to use a REDCap database for data collection and monitoring. Patient specific data will be entered by study personnel into the REDCap database after completion of the patient's intervention and postoperative followup. This will avoid disrupting the blinding of study personnel gathering postoperative pain data. Postoperative narcotic use will be gathered from a chart review of ordered and administered medications.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or older
* low energy mechanism (i.e. mechanical or syncopal fall from ground level)
* extracapsular location as defined on AP and lateral radiographs of the hip

Exclusion Criteria:

* polytrauma patients with multiple injuries, high energy mechanisms (i.e. pedestrian struck, motor vehicle collision, fall from height)
* inability for the patient to consent for themselves
* pathologic fracture types (secondary to tumor or atypical fractures due to bisphosphonate use)
* intolerance or allergies to opioids or local anesthetics

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scores | 24 hours
  The pain visual analog scale will be used to record pain scores from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Opioid usage | 24 hours
  The amount of opioid pain medications used in the 24-hour postoperative period will be converted to morphine equivalents as published by the Center for Medicare and Medicaid Services and summed.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sen, Principal Investigator — Jacobi Medical Center; Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnea R, Weiss Y, Abadi-Korek I, Shemer J. The epidemiology and economic burden of hip fractures in Israel. Isr J Health Policy Res. 2018 Aug 2;7(1):38. doi: 10.1186/s13584-018-0235-y. PMID 30068383
- [Background] Sadat-Ali M, Alfaraidy M, AlHawas A, Al-Othman AA, Al-Dakheel DA, Tayara BK. Morbidity and mortality after fragility hip fracture in a Saudi Arabian population: Report from a single center. J Int Med Res. 2017 Jun;45(3):1175-1180. doi: 10.1177/0300060517706283. Epub 2017 May 8. PMID 28480812
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Malik AT, Quatman CE, Phieffer LS, Ly TV, Khan SN. Incidence, risk factors and clinical impact of postoperative delirium following open reduction and internal fixation (ORIF) for hip fractures: an analysis of 7859 patients from the ACS-NSQIP hip fracture procedure targeted database. Eur J Orthop Surg Traumatol. 2019 Feb;29(2):435-446. doi: 10.1007/s00590-018-2308-6. Epub 2018 Sep 18. PMID 30229446
- [Background] Sieber FE, Mears S, Lee H, Gottschalk A. Postoperative opioid consumption and its relationship to cognitive function in older adults with hip fracture. J Am Geriatr Soc. 2011 Dec;59(12):2256-62. doi: 10.1111/j.1532-5415.2011.03729.x. Epub 2011 Nov 7. PMID 22092232
- [Background] Morrison SR, Magaziner J, McLaughlin MA, Orosz G, Silberzweig SB, Koval KJ, Siu AL. The impact of post-operative pain on outcomes following hip fracture. Pain. 2003 Jun;103(3):303-311. doi: 10.1016/S0304-3959(02)00458-X. PMID 12791436
- [Background] Amin NH, West JA, Farmer T, Basmajian HG. Nerve Blocks in the Geriatric Patient With Hip Fracture: A Review of the Current Literature and Relevant Neuroanatomy. Geriatr Orthop Surg Rehabil. 2017 Dec;8(4):268-275. doi: 10.1177/2151458517734046. Epub 2017 Oct 13. PMID 29318091
- [Background] Swenson JD, Davis JJ, Stream JO, Crim JR, Burks RT, Greis PE. Local anesthetic injection deep to the fascia iliaca at the level of the inguinal ligament: the pattern of distribution and effects on the obturator nerve. J Clin Anesth. 2015 Dec;27(8):652-7. doi: 10.1016/j.jclinane.2015.07.001. Epub 2015 Aug 13. PMID 26277873
- [Background] Steenberg J, Moller AM. Systematic review of the effects of fascia iliaca compartment block on hip fracture patients before operation. Br J Anaesth. 2018 Jun;120(6):1368-1380. doi: 10.1016/j.bja.2017.12.042. Epub 2018 Apr 5. PMID 29793602
- [Background] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Background] Dickman E, Pushkar I, Likourezos A, Todd K, Hwang U, Akhter S, Morrison S. Ultrasound-guided nerve blocks for intracapsular and extracapsular hip fractures. Am J Emerg Med. 2016 Mar;34(3):586-9. doi: 10.1016/j.ajem.2015.12.016. Epub 2015 Dec 14. PMID 26809928
- [Background] Li J, Dai F, Chang D, Harmon E, Ibe I, Sukumar N, Halaszynski TM, Rubin LE, O'Connor MI. A Practical Analgesia Approach to Fragility Hip Fracture: A Single-Center, Retrospective, Cohort Study on Femoral Nerve Block. J Orthop Trauma. 2019 Apr;33(4):175-179. doi: 10.1097/BOT.0000000000001391. PMID 30570615
- [Background] Madabushi R, Rajappa GC, Thammanna PP, Iyer SS. Fascia iliaca block vs intravenous fentanyl as an analgesic technique before positioning for spinal anesthesia in patients undergoing surgery for femur fractures-a randomized trial. J Clin Anesth. 2016 Dec;35:398-403. doi: 10.1016/j.jclinane.2016.09.014. Epub 2016 Oct 14. PMID 27871563
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Background] Mangram AJ, Oguntodu OF, Hollingworth AK, Prokuski L, Steinstra A, Collins M, Sucher JF, Ali-Osman F, Dzandu JK. Geriatric trauma G-60 falls with hip fractures: A pilot study of acute pain management using femoral nerve fascia iliac blocks. J Trauma Acute Care Surg. 2015 Dec;79(6):1067-72; discussion 1072. doi: 10.1097/TA.0000000000000841. PMID 26680143
- [Background] Singh GK, Manglik RK, Lakhtakia PK, Singh A. Analgesia for the reduction of Colles fracture. A comparison of hematoma block and intravenous sedation. Online J Curr Clin Trials. 1992 Oct 1;Doc No 23:[3614 words; 43 paragraphs]. PMID 1343612
- [Background] White BJ, Walsh M, Egol KA, Tejwani NC. Intra-articular block compared with conscious sedation for closed reduction of ankle fracture-dislocations. A prospective randomized trial. J Bone Joint Surg Am. 2008 Apr;90(4):731-4. doi: 10.2106/JBJS.G.00733. PMID 18381308